CLINICAL TRIAL: NCT03171454
Title: Randomized, Controlled Trial Comparing Immediate and Delayed Intrauterine Balloon Therapy in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Brief Title: Immediate and Delayed Intrauterine Balloon in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoyu Shi, Principal Investigator, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017FXHEC-KY006
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Intrauterine Adhesion
Keywords: hysteroscopic operation; intrauterine balloon; adhesions
MeSH Terms: conditions — Gynatresia; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Intrauterine Balloon therapy (Experimental): In the delayed balloon group,a Foley catheter will be inserted into the uterine cavity 2 weeks after the surgery, the balloon will be inflated with normal saline (from 3ml to 5ml) then deflated, and the procedure repeated three time over 3 minutes or so, then the cavity will be flushed with 10 mls of normal saline solution after via the irrigating channel of the Foley catheter before removal. The whole procedure will be repeated a further 2 weeks later.
  Interventions: Procedure: Delayed Intrauterine Balloon therapy
- immediate Intrauterine Balloon therapy (Experimental): At the conclusion of the surgery, in the immediate balloon group: a Foley-catheter will be immediately inserted into the uterine cavity and the balloon will be distended with 5mls of saline under ultrasound guidance and the balloon will stay in situ for 7 days.
  Interventions: Procedure: immediate Intrauterine Balloon therapy

INTERVENTIONS:
Procedure: Delayed Intrauterine Balloon therapy — D-IUB dilatation therapy group will be performed using a (size 12-14fr) Foley catheter and according to the methodology published in the literature. This will be prepared by cutting the catheter tip protruding beyond the balloon. Once the catheter has reached the fundus, 5mls of saline will be slowly instilled into the balloon under ultrasound guidance.
  Arms: Delayed Intrauterine Balloon therapy
Procedure: immediate Intrauterine Balloon therapy — At the conclusion of the surgery, in the immediate balloon group: a Foley-catheter will be immediately inserted into the uterine cavity and the balloon will be distended with 4-5mls of saline under ultrasound guidance and the balloon will stay in situ for 7 days.
  Arms: immediate Intrauterine Balloon therapy

SUMMARY:
In this prospective, randomized, controlled study, the investigators wish to compare the efficacy of immediate and delayed intrauterine balloon (IUB) therapy in the prevention of adhesion reformation after hysteroscopic adhesiolysis.

DETAILED DESCRIPTION:
Objectives

To compare the efficacy of placing an Intrauterine Balloon immediately after surgery and delayed Intrauterine Balloon Dilatation Therapy after surgery in the prevention of adhesion reformation after hysteroscopic adhesiolysis.

Patients

The patients will be recruited from two centers, namely, the HysterscopyCenter of the Fuxing Hospital and TianTan Hospital, Capital Medical University, Beijing, China.Before the surgery all patients with suspected Asherman syndrome will undergo preoperative evaluations, including a detailed history of the menstrual pattern, any previous intrauterine surgery, and reproductive history, as well as trans-vaginal ultrasonography.The severity and extent of intrauterine adhesions will be scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version). The inclusion criteria include [1] women aged 18-40 years; [2] moderate to severe intrauterine adhesion (AFS score≥5); [3] first episode of hysteroscopic adhesiolysis in the investigators hospital; [4] written consent obtained; and [5] agreement to have second-look hysteroscopy. The exclusion criteria include [1] minimal adhesion (AFS score <5) and [2] previous hysteroscopic adhesiolysis in the investigators hospital.

Study Design

At the conclusion of hysteroscopic adhesiolysis, recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: [1] Immediate Intrauterine Balloon therapy (I-IUB) group: Immediately place a Foley-catheter intrauterine balloon which will be removed after 7 days after surgery; [2] Delayed Intrauterine Balloon therapy (D-IUB) group： insertion of a Foley-catheter to distend the uterine cavity 2 weeks and 4 weeks after hysteroscopic adhesiolysis; A second-look hysteroscopy will be carried out in the early proliferative phase 6 weeks after the surgery.

Power Calculation

On the basis of the results of the two published retrospective cohort studies comparing the balloon and hormone therapy group (control group) in the prevention of adhesion reformation, the investigators estimate that the adhesion reformation rate in the immediate balloon group to be 30% and in the delayed balloon group to be 10%. Accepting a type 1 error of 0.05, and a type 2 error of 0.10, the number of subjects in each arm of the randomized, controlled trial would be 79. Assuming that the dropout rate to be 20%, the total number of subject to be recruited would be 90 in each arm.

Procedure

Surgical procedure

The surgery will be carried out by one of three experienced hysteroscopic surgeons with the use of a 8.5-mm rigid hysteroscope (Olympus) with 0.9% normal saline infusion under 100-120 mmHg pressure. The procedure will be performed under general anesthesia in a day surgery unit. Ultrasonographic guidance will be routinely used. Once the extent and severity of uterine adhesion has been assessed, the adhesions will be divided with the use of bipolar instrument until normal uterine anatomy is achieved.At the conclusion of the surgery, in the immediate balloon group: a Foley-catheter will be immediately inserted into the uterine cavity and the balloon will be distended with 5mls of saline under ultrasound guidance and the balloon will stay in situ for 7 days. In the delayed balloon group,a Foley catheter will be inserted into the uterine cavity 2 weeks after the surgery, the balloon will be inflated with normal saline (from 3-5ml) then deflated, and the procedure repeated three time over 3 minutes or so, then the cavity will be flushed with 10 mls of normal saline solution after via the irrigating channel of the Foley catheter before removal. The whole procedure will be repeated a further 2 weeks later.

Postoperative treatments

All subjects will be treated with oral antibiotics for 5 days. In all cases hormone therapy will also begin from the day of operation, consisting of estradiol at a dose of 2 mg, bid for 21- 28 days, with the addition of dydrogesterone at a dose of 10 mg, bid for the last 10 days of the estrogen therapy. After the withdrawal bleed, the hormone therapy will be repeated for another cycle. Second-look hysteroscopy will be carried out in the early proliferative phase, 6 weeks after the initial operation. After assessment of the extent and severity of any reformed adhesion, hysteroscopic adhesiolysis will also be carried out at the time of the second-look procedure, if adhesion has recurred. The surgeon who performs the second-look hysteroscopy will be blinded to the randomization.

IUB dilatation

D-IUB dilatation therapy group will be performed using a Foley catheter and according to the methodology published in the literature. This will be prepared by cutting the catheter tip protruding beyond the balloon. Once the catheter has reached the fundus, 5mls of saline will be slowly instilled into the balloon under ultrasound guidance.

Statistical Analysis

The rate of the recurrence of adhesion in the two groups will be compared using the χ2 test. The reduction of AFS score in the two groups will be compared using the Mann-Whitney U test. A p value of < 0.05 will be considered statistically significant. All statistical analysis will be carried out with the use of SPSS 21.0.

Outcome measures

The primary outcome measure will include the degree of intrauterine adhesions and AFS score at follow-up. The secondary outcome measures will include the change of menstrual pattern after surgery and the need for re-operation.The third outcome measures will include any complications including any clinicalinfection.

Data processing and analysis

The researchers will ensure the confidentiality of sensitive data by minimizing the number of personnel who handle subject data. In addition, computer data will be encrypted as required to maximize security, while paper documents will be locked in filing cabinets, with only authorized personnel having access to the information.

Ethical considerations

IUB dilatation has been published as a novel technique with no untoward complications identified to date. The procedure will be performed according to the methodology available in the literature and the study has gained approval from the local ethical committee.

Consent

All subjects will be given a detailed explanation of the study and sufficient time to consider participants. A written consent form will be signed by the patient and retained in the investigators confidential records

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-40 years;
* moderate to severe intrauterine adhesion (AFS score≥5);
* first episode of hysteroscopicadhesiolysis in our hospital;
* written consent obtained;
* agreement to have second-look hysteroscopy.

Exclusion Criteria:

* minimal adhesion (AFS score <5)
* previous hysteroscopic adhesiolysis in our hospital.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
AFS score | at 6 weeks post-op
  The degree of intrauterine adhesions described by AFS score reduction at second look hysteroscopy

SECONDARY OUTCOMES:
The menstrual pattern | at 6 weeks post-op
  Menstrual blood loss figure before and after surgery
infection rate | at 6 weeks post-op
  Secretion bacteria culture

CONTACTS AND LOCATIONS:
Overall Officials: Tinchiu Li, Study Chair — Fu Xing Hospital, Capital Medical University
Locations (1):
- Fu Xing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] March CM. Intrauterine adhesions. Obstet Gynecol Clin North Am. 1995 Sep;22(3):491-505. PMID 8524533
- [Result] Saravelos SH, Li TC. Ultrasound-guided treatment of intrauterine adhesions in the outpatient setting. Ultrasound Obstet Gynecol. 2017 Aug;50(2):278-280. doi: 10.1002/uog.16218. No abstract available. PMID 27420903
- [Result] Saravelos SH and Li TC. Intrauterine balloon therapy: a novel ultrasound guided treatment for intrauterine adhesions. Gynecological Surgery [Epub ahead of print]
- [Result] Saravelos SH, Jayaprakasan K, Ojha K, Li TC. Assessment of the uterus with three-dimensional ultrasound in women undergoing ART. Hum Reprod Update. 2017 Mar 1;23(2):188-210. doi: 10.1093/humupd/dmw040. PMID 28007752
- [Result] Orhue AA, Aziken ME, Igbefoh JO. A comparison of two adjunctive treatments for intrauterine adhesions following lysis. Int J Gynaecol Obstet. 2003 Jul;82(1):49-56. doi: 10.1016/s0020-7292(03)00030-4. PMID 12834941
- [Result] Taskin O, Sadik S, Onoglu A, Gokdeniz R, Erturan E, Burak F, Wheeler JM. Role of endometrial suppression on the frequency of intrauterine adhesions after resectoscopic surgery. J Am Assoc Gynecol Laparosc. 2000 Aug;7(3):351-4. doi: 10.1016/s1074-3804(05)60478-1. PMID 10924629
- [Result] Healy MW, Schexnayder B, Connell MT, Terry N, DeCherney AH, Csokmay JM, Yauger BJ, Hill MJ. Intrauterine adhesion prevention after hysteroscopy: a systematic review and meta-analysis. Am J Obstet Gynecol. 2016 Sep;215(3):267-275.e7. doi: 10.1016/j.ajog.2016.05.001. Epub 2016 May 10. PMID 27173082
- [Result] Guida M, Acunzo G, Di Spiezio Sardo A, Bifulco G, Piccoli R, Pellicano M, Cerrota G, Cirillo D, Nappi C. Effectiveness of auto-crosslinked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic surgery: a prospective, randomized, controlled study. Hum Reprod. 2004 Jun;19(6):1461-4. doi: 10.1093/humrep/deh238. Epub 2004 Apr 22. PMID 15105384
- [Result] Roge P, D'Ercole C, Cravello L, Boubli L, Blanc B. Hysteroscopic management of uterine synechiae: a series of 102 observations. Eur J Obstet Gynecol Reprod Biol. 1996 Apr;65(2):189-93. doi: 10.1016/0301-2115(95)02342-9. PMID 8730623
- [Result] Schenker JG. Etiology of and therapeutic approach to synechia uteri. Eur J Obstet Gynecol Reprod Biol. 1996 Mar;65(1):109-13. doi: 10.1016/0028-2243(95)02315-j. PMID 8706941
- [Result] Pabuccu R, Atay V, Orhon E, Urman B, Ergun A. Hysteroscopic treatment of intrauterine adhesions is safe and effective in the restoration of normal menstruation and fertility. Fertil Steril. 1997 Dec;68(6):1141-3. doi: 10.1016/s0015-0282(97)00375-0. PMID 9418714